# INFORMATIE VOOR PATIËNTEN EN VERKLARING VAN BEREIDHEID TOT DEELNAME

# COVID-19: Een studie over aerosolvorming tijdens een gastroscopie (endoscopisch maagonderzoek) met een aangepast mondstuk voor druppelvermindering

I-Hsuan Huang, Pieter Sinonquel, Kristof Buysschaert, Hilde Willekens, Herman Devriese, Raf Bisschops & Jan Tack

| Registratie nummer: S65197 | |
|------------------------------------|-------------------------|
| (toegekend door Ethische Commissie | Onderzoek UZ/KU Leuven) |

# Onderzoeksinstelling:

- Translational Research Center for Gastrointestinal Disorders (TARGID), Katholieke Universiteit (KU) Leuven
- Universitair Ziekenhuis (UZ) Gasthuisberg, Leuven, Belgium

Principal investigator: Prof. Dr. Jan Tack

University Hospital Gasthuisberg Katholieke Universiteit Leuven

Herestraat 49 - bus 701

B-3000 Leuven

# I Noodzakelijke informatie voor uw beslissing om deel te nemen

# Inleiding

Voordat u beslist over uw deelname aan deze studie willen we u wat meer informatie geven over wat dit betekent op organisatorisch vlak en wat de eventuele voordelen en risico's voor u zijn. Zo kan u een beslissing nemen op basis van de juiste informatie. Dit wordt "geïnformeerde toestemming" genoemd.

Wij vragen u de volgende pagina's met informatie aandachtig te lezen. Hebt u vragen, dan kan u terecht bij de arts-onderzoeker of zijn vertegenwoordiger. Dit document bestaat uit 3 delen: essentiële informatie die u nodig heeft voor het nemen van uw beslissing, uw schriftelijke toestemming en bijlagen waarin u meer details terug kan vinden over bepaalde onderdelen van de basisinformatie.

Als u aan deze klinische studie deelneemt, dient u het volgende te weten:

- De klinische studie wordt opgestart na evaluatie door de Ethische Commissie
   Onderzoek UZ/KU Leuven.
- Uw deelname is vrijwillig; er kan op geen enkele manier sprake zijn van dwang. Voor deelname is uw ondertekende toestemming nodig. Ook nadat u hebt getekend, kan u de arts-onderzoeker laten weten dat u uw deelname wilt stopzetten. De beslissing om al dan niet (verder) deel te nemen zal geen enkele negatieve invloed hebben op de kwaliteit van de zorgen noch op de relatie met de behandelende arts(en).
- De gegevens die in het kader van uw deelname worden verzameld, zijn vertrouwelijk. Bij de publicatie van de resultaten is uw anonimiteit verzekerd.
- Er worden u geen kosten aangerekend voor specifieke behandelingen, bezoeken of consultaties, onderzoeken in het kader van deze studie.
- Er is een verzekering afgesloten voor het geval dat u schade zou oplopen in het kader van uw deelname aan deze klinische studie.
- Indien u extra informatie wenst, kan u altijd contact opnemen met de artsonderzoeker of een medewerker van zijn team.
- Wij raden aan uw huisarts op de hoogte te brengen wanneer u deelneemt aan een klinische studie.

Aanvullende informatie over "Rechten van de deelnemer aan een klinische studie" vindt u in bijlage pagina 9.

# Achtergrond en doel van de studie

Tijdens onderzoeken op de endoscopie eenheid gaat men na hoe het maag- en darmstelsel functioneert. Om het maag- en darmstelsel te onderzoeken gebruikt men vaak een endoscoop. Dit is een flexibele buis met een camera die de slokdarm, maag en het begin van de dunne darm (duodenum) in beeld kan brengen tijdens een endoscopisch maagonderzoek (gastroscopie). Tijdens een gastroscopie kunnen kleine (speeksel)druppeltjes van de patiënt in de lucht terechtkomen door de ingeblazen lucht en ook bij kuchen, hoesten, braken, etc. Uit eerder wetenschappelijk onderzoek is bovendien gebleken dat deze kleine druppeltjes wel tot 3 uur in de lucht blijven circuleren en nadien kunnen neerdalen op oppervlakten in de onderzoeksruimte.

Indien die druppeltjes afkomstig zijn van een patiënt met een virale luchtweginfectie is het mogelijk dat zij een hoge virale lading bevatten, wat wil zeggen dat er veel (besmettelijke) ziektekiemen aanwezig kunnen zijn in deze druppeltjes. Uit wetenschappelijk onderzoek is gebleken dat er bij mensen met virale infecties in deze regio (neus-, keel-, en mondholte) ook een hoog aantal (besmettelijke) ziektekiemen aanwezig zijn. Gezondheidsmedewerkers werkzaam op de 'Functiemetingen endoscopie' eenheid kunnen dus een verhoogd risico hebben op verschillende infectieziekten doordat zij dagelijks dergelijke onderzoeken uitvoeren.

Tijdens de coronapandemie is het risico van gezondheidsmedewerkers werkzaam op de endoscopie eenheid opnieuw bevestigd, waardoor verschillende centra in Europa hebben besloten om hun werkcapaciteit met 50 – 100 % te verminderen. Op dit moment bevinden we ons in de nasleep van de corona pandemie waarbij er beschermingsmaatregelen worden genomen om zowel patiënten als personeel te beschermen tegen de verdere verspreiding van het coronavirus. Patiënten worden voorafgaand aan hun onderzoek getest om een mogelijke besmetting met het coronavirus op te sporen en in het ziekenhuis is het dragen van een mondmasker verplicht. Personeel op de endoscopie eenheid draagt een mondmasker, handschoenen, beschermingsbril, haarnet en een waterbestendige schort. Tijdens een gastroscopie is het voor een patiënt niet mogelijk om een mondmasker op te houden omdat de scoop (flexibele buis) via de mond moet worden binnengebracht. Om te vermijden dat er wordt gebeten op de scoop, wordt er steeds een mondstuk tussen de tanden van de patiënt geplaatst. Er werd recent een speciaal mondstuk ontwikkeld dat druppelverspreiding zou verminderen. Dit mondstuk heeft een ingebouwd sponsstukje dat de opening wat meer afsluit, en een bijkomende plaat in doorzichtig buigzaam plastiek die druppeltjes moet tegenhouden.

Daar er een tekort is aan wetenschappelijk onderzoek over de hoeveelheid en de spreiding van de (speeksel)druppeltjes tijdens een maagonderzoek, willen wij deze hoeveelheid en verspreiding van (speeksel)druppeltjes meten tijdens onderzoeken waarbij we het standaard mondstuk of het meer afgesloten mondstuk gebruiken. Beide mondstukken zijn op de markt in België en voldoen aan alle regels en vereisten voor een medisch hulpmiddel.

# Verloop van de studie

U komt in aanmerking voor deze studie omdat bij u een gastroscopie gepland is. Graag geven we u wat meer informatie over het verloop van dit onderzoek.

Eén of maximum twee dagen voorafgaand aan uw gepland maagonderzoek, zal u een wisser krijgen om na te gaan of u besmet bent met Covid-19. Het maagonderzoek kan enkel plaatsvinden bij een negatief testresultaat van deze wisser.

Op de dag van uw gastroscopie wordt u nuchter verwacht. U kan kiezen of dit maagonderzoek al dan niet onder verdoving (roesje) gebeurt. Bij iedereen wordt er wat plaatselijke verdoving (xylocaïne spray) in de keel gespoten om de kokhalsreflex te verminderen.

Wanneer u beslist om deel te nemen aan deze studie, zijn er twee zaken, die hieronder worden opgesomd, die anders zullen verlopen dan wanneer u niet deelneemt aan deze studie.

- Bij deelname aan de studie zal er via loting worden bepaald of er tijdens uw onderzoek zal worden gebruik gemaakt van het standaardmondstuk of van het nieuw ontwikkelde mondstuk. Het nieuwe mondstuk is wat nauwer afgesloten rond de scoop en is omrand met een soepel plastiek scherm (zie afbeelding)
- er vlak voor, na en tijdens de gastroscopie met een deeltjesteller worden gemeten hoeveel partikels en druppeltjes er in de lucht van de onderzoeksruimte aanwezig zijn. De meting zal gebeuren 1, 3, 5, 10 en 15 minuten na start van de gastroscopie en vlak nadat de scoop wordt verwijderd. Het is mogelijk dat er geen telling na 10 en/of 15 minuten zal plaatsvinden, indien uw onderzoek reeds vroeger werd beëindigd. Een deeltjesteller is een draagbaar apparaat dat wordt vastgehouden door een persoon die naast de onderzoekstafel staat. U ondervindt hiervan zelf geen enkele hinder.



## Kan ik deelnemen aan de studie?

Voor deze studie zijn we op zoek naar mannen en vrouwen ouder dan 18 jaar bij wie reeds een gastroscopie gepland is.

U kan niet deelnemen indien u zwanger bent of borstvoeding geeft.

# Contact

Als u bijkomende informatie wenst, maar ook ingeval van problemen of als u zich zorgen maakt, kan u contact opnemen met de arts-onderzoeker (Prof. Dr. Jan Tack) of een medewerker van zijn studieteam:

Prof. Dr. Jan Tack op het telefoonnummer 016/34.42.25

Hilde Willekens op het telefoonnummer 016/34.03.96

Lieselot Holvoet op het telefoonnummer 016/34.07.50

Als u vragen hebt met betrekking tot uw rechten als deelnemer aan de studie, kan u contact opnemen met de ombudsdienst in uw ziekenhuis op het telefoonnummer: 016/34.48.18. Indien nodig kan de ombudsdienst u in contact brengen met het Ethisch Comité.

Een studie over aerosol verspreiding tijdens gastro-intestinale motiliteits onderzoeken

## II Geïnformeerde toestemming

Ik verklaar dat ik geïnformeerd ben over de aard, het doel, de duur, de eventuele voordelen en risico's van de studie en dat ik weet wat van mij wordt verwacht. Ik heb kennisgenomen van het informatiedocument en de bijlagen ervan.

Ik heb voldoende tijd gehad om na te denken en met een door mij gekozen persoon, zoals mijn huisarts of een familielid, te praten.

Ik heb alle vragen kunnen stellen die bij me opkwamen en ik heb een duidelijk antwoord gekregen op mijn vragen.

Ik begrijp dat mijn deelname aan deze studie vrijwillig is en dat ik vrij ben mijn deelname aan deze studie stop te zetten zonder dat dit mijn relatie schaadt met het therapeutisch team dat instaat voor mijn gezondheid.

Ik begrijp dat er tijdens mijn deelname aan deze studie gegevens over mij zullen worden verzameld en dat de arts-onderzoeker en de opdrachtgever de vertrouwelijkheid van deze gegevens verzekeren overeenkomstig de Europese en Belgische wetgeving ter zake. Ik begrijp dat het uitvoeren van deze studie door UZ Leuven het algemeen belang dient en de verwerking van mijn persoonsgegevens noodzakelijk is voor het uitvoeren van deze studie.

Ik heb een exemplaar ontvangen van de informatie aan de deelnemer en de geïnformeerde toestemming.

Naam en voornaam:

Datum:

Handtekening van de deelnemer:

#### **Arts-onderzoeker**

Ik, ondergetekende arts-onderzoeker, verklaar de benodigde informatie inzake deze studie mondeling te hebben verstrekt evenals een exemplaar van het informatiedocument aan de deelnemer te hebben verstrekt.

Ik bevestig dat geen enkele druk op de deelnemer is uitgeoefend om hem/haar te doen toestemmen tot deelname aan de studie en ik ben bereid om op alle eventuele bijkomende vragen te antwoorden.

Ik bevestig dat ik werk in overeenstemming met de ethische beginselen zoals vermeld in de laatste versie van de "Verklaring van Helsinki", de "Goede klinische praktijk" en de Belgische wet van 7 mei 2004 inzake experimenten op de menselijke persoon.

Datum:

Handtekening:

Een studie over aerosolvorming tijdens een gastroscopie (endoscopisch maagonderzoek) met een aangepast mondstuk voor druppelvermindering

#### III Aanvullende informatie

# Aanvullende informatie over de risico's die verbonden zijn aan de deelname aan deze studie

De onderzoeken die in deze studie worden verricht brengen geen of slechts een zeer gering en voorspelbaar risico met zich mee.

De dagen na een gastroscopie kan u een beetje last hebben van keelpijn. Wanneer u verdoving (roesje) kreeg tijdens het onderzoek, kan u zich nadien een beetje suf voelen en mag u die dag niet meer zelf met de auto rijden.

# Aanvullende informatie over de bescherming en de rechten van de deelnemer aan een klinische studie

# Ethisch comité

Deze studie werd geëvalueerd door een onafhankelijk ethisch comité, de Ethische Commissie Onderzoek UZ/KU Leuven, die een gunstig advies heeft uitgebracht. De ethische comités hebben als taak de personen die aan klinische studies deelnemen te beschermen. Ze controleren of uw rechten als patiënt en als deelnemer aan een studie gerespecteerd worden, of de studie wetenschappelijk relevant en ethisch verantwoord is.

Hierover brengen de ethische comités een advies uit in overeenstemming met de Belgische wet van 7 mei 2004.

U dient het positief advies van de Ethische Comités in geen geval te beschouwen als een aansporing om deel te nemen aan deze studie.

# Vrijwillige deelname

Aarzel niet om alle vragen te stellen die u nuttig vindt voordat u tekent. Neem de tijd om er met een vertrouwenspersoon over te praten, als u dit wenst.

U heeft het recht om niet deel te nemen aan deze studie of met deze studie te stoppen zonder dat u hiervoor een reden hoeft te geven, zelfs al hebt u eerder toegestemd om aan deze studie deel te nemen. Uw beslissing zal in geen geval uw relatie met de artsonderzoeker en de voortzetting van uw therapeutische behandeling veranderen.

Als u aanvaardt om aan deze studie deel te nemen, ondertekent u het toestemmingsformulier. De arts-onderzoeker zal dit formulier ook ondertekenen en zal zo

bevestigen dat hij u de noodzakelijke informatie voor deze studie heeft gegeven. U zult het voor u bestemde exemplaar ontvangen.

## Kosten in verband met uw deelname

Uw deelname zal voor u geen bijkomende kosten met zich meebrengen. In deze studie, verbonden aan een onderzoek dat voor uw gezondheidstoestand uitgevoerd wordt, is geen vergoeding voor uw deelname voorzien.

#### Voordelen en vergoedingen

Deelname aan deze studie zal u geen direct voordeel opleveren. Wij hopen dat de resultaten bekomen uit deze studie zullen kunnen bijdragen tot een beter begrip van de spreiding van partikels tijdens maagonderzoeken.

## Vertrouwelijkheidgarantie

Uw deelname aan de studie betekent dat de arts-onderzoeker gegevens over u verzamelt en dat de opdrachtgever van de studie die gebruikt voor onderzoek en in het kader van wetenschappelijke en medische publicaties. De verwerking van uw persoonsgegevens is noodzakelijk om de wetenschappelijke onderzoeksdoeleinden zoals hierin te kunnen realiseren. Het uitvoeren van academische onderzoek behoort tot wettelijke opdrachten van UZ Leuven als opdrachtgever. Als universitair ziekenhuis verbonden aan de KU Leuven dient UZ Leuven immers wetenschap en onderwijs in het algemeen belang te ondersteunen. UZ Leuven verduidelijkt u graag dat de noodzakelijkheid van de verwerking voor het uitvoeren van wetenschappelijk onderzoek en dit als taak van algemeen belang, de wettelijke toelatingsgrond vormt op basis waarvan UZ Leuven in het kader van dit onderzoek uw gegevens verwerkt. Daarnaast is UZ Leuven onderhevig aan specifieke wettelijke verplichtingen die de verwerking van uw gegevens mogelijks noodzakelijk maken in het kader van veiligheidsrapportering (zoals bijvoorbeeld het melden van bijwerkingen aan toezichthoudende overheidsinstanties).

Uw gegevens zullen worden verwerkt overeenkomstig de Europese Algemene Verordening inzake Gegevensbescherming (AVG) en de Belgische Wetgeving betreffende de bescherming van natuurlijke personen met betrekking tot de verwerking van persoonsgegevens. KULeuven – UZ Leuven is de verwerkingsverantwoordelijke voor uw gegevens.

U hebt het recht om aan de arts-onderzoeker te vragen welke gegevens hij/zij over u heeft verzameld en waarvoor ze gebruikt worden in het kader van de studie. Deze gegevens hebben betrekking op uw huidige klinische situatie maar ook op uw medische voorgeschiedenis en op de resultaten van onderzoeken die werden uitgevoerd voor de

behandeling van uw gezondheid volgens de geldende zorgstandaard. U hebt het recht om deze gegevens in te kijken en om verbeteringen te laten aanbrengen indien ze foutief zouden zijn<sup>1</sup>.

De arts-onderzoeker is verplicht om deze verzamelde gegevens vertrouwelijk te behandelen.

Dit betekent dat hij zich ertoe verbindt om uw naam nooit bekend te maken in het kader van een publicatie of een conferentie en dat hij uw gegevens zal coderen (uw identiteit zal worden vervangen door een identificatiecode in de studie) voordat hij ze doorgeeft aan de beheerder van de databank (KULeuven – TARGID – Herestraat 49 bus 701 – 3000 Leuven).

De arts-onderzoeker en zijn team zullen gedurende de volledige klinische studie de enige personen zijn die een verband kunnen leggen tussen de overgedragen gegevens en uw medisch dossier <sup>2</sup>.

De overgedragen persoonlijke gegevens omvatten geen combinatie van elementen waarmee het mogelijk is u te identificeren <sup>3</sup>.

De door de opdrachtgever aangestelde beheerder van de onderzoeksgegevens kan u niet identificeren op basis van de overgedragen gegevens. Deze persoon is verantwoordelijk voor het verzamelen van de gegevens die door alle artsen-onderzoekers die deelnemen aan de studie zijn verzameld en voor de verwerking en de bescherming van die gegevens in overeenstemming met de Belgische wet betreffende de bescherming van de persoonlijke levenssfeer.

Om de kwaliteit van de studie te controleren, kan uw medisch dossier worden ingekeken door personen die gebonden zijn aan het beroepsgeheim zoals vertegenwoordigers van de ethische comités, van de opdrachtgever van de studie of een extern auditbureau. Dit kan enkel gebeuren onder strikte voorwaarden, onder de verantwoordelijkheid van de artsonderzoeker en onder zijn/haar toezicht (of van één van zijn/haar onderzoeksmedewerkers).

Uw toestemming om aan deze studie deel te nemen betekent dat uw gecodeerde medische gegevens gebruikt worden voor doeleinden die in dit informatieformulier staan beschreven en dat ze worden overgedragen aan bovenvermelde personen en/of instellingen.

De opdrachtgever verbindt zich ertoe om de verzamelde gegevens enkel in het kader van deze studie te gebruiken.

3 De database met de resultaten van de studie zal dus geen elementen bevatten zoals uw initialen, uw geslacht en uw volledige geboortedatum (dd/mm/jijj).

Informatie- en toestemmingsdocument Aerosolvorming tijdens gastroscopie (S65197) versie 2, 02/03/2021

<sup>1</sup> Deze rechten zijn bepaald door de Europese Algemene Verordening Gegevensbescherming (AVG), door de Belgische Wetgeving betreffende de bescherming van natuurlijke personen met betrekking tot de verwerking van persoonsgegevens en door de wet van 22 augustus 2002 betreffende de rechten van de patiënt.

<sup>&</sup>lt;sup>2</sup> De wet verplicht om voor klinische studies dit verband met uw dossier gedurende 20 jaar te bewaren.

Indien u uw toestemming tot deelname aan de studie intrekt, zullen de gecodeerde gegevens

die al verzameld waren vóór uw terugtrekking, bewaard worden. Hierdoor wordt de

geldigheid van de studie gegarandeerd. Er zal geen enkel nieuw gegeven aan de

opdrachtgever worden doorgegeven.

Indien u vragen hebt over hoe wij uw gegevens gebruiken, dan kan u hiervoor steeds terecht

bij uw arts-onderzoeker. Ook de functionaris voor gegevensbescherming van het

onderzoekcentrum staan ter uwer beschikking.

De contactgegevens van deze laatste zijn als volgt: DPO - UZ Leuven, Herestraat 49, 3000

Leuven, e-mail dpo@uzleuven.be.

Tot slot, indien u een klacht heeft over de verwerking van uw gegevens, kunt u contact

opnemen met de Belgische toezichthoudende instantie die toeziet op de naleving van de

grondbeginselen van de bescherming van persoonsgegevens:

De Belgische toezichthoudende instantie heet:

Gegevensbeschermingsautoriteit (GBA)

Drukpersstraat 35,

1000 Brussel

Tel. +32 2 274 48 00

e-mail: contact(at)apd-gba.be

Website: http://www.gegevensbeschermingsautoriteit.be

Verzekering

Voor deze studie heeft de opdrachtgever, UZ Leuven, een verzekering afgesloten met

Contractnummer 299.053.700. De studie is verzekerd in overeenstemming met de

bepalingen van art.29 van de Belgische wet van 07/05/2004 inzake experimenten op de

menselijke persoon.

Elke deelname aan een studie houdt een risico in, hoe klein ook. De opdrachtgever is - ook

indien er geen sprake is van fout - aansprakelijk voor de schade die de deelnemer of in geval

van overlijden zijn/haar rechthebbenden, oplopen en die rechtstreeks of onrechtstreeks

verband houdt met diens deelname aan de studie. De opdrachtgever heeft voor deze

aansprakelijkheid een verzekering afgesloten.

We verzoeken u daarom om elk nieuw gezondheidsprobleem aan de arts-onderzoeker te

melden alvorens een andere arts te raadplegen, een (ander) geneesmiddel in te nemen of

een andere medische behandeling te ondergaan. Indien u om eender welke reden

gedurende deze klinische studie een andere arts raadpleegt, dient u deze te melden dat u deelneemt aan een klinische studie. Dit kan belangrijk zijn voor een juiste diagnose en behandeling van uw klachten.

Indien de arts-onderzoeker van mening is dat er een verband met de studie mogelijk is, zal hij/zij de opdrachtgever van de studie op de hoogte stellen die de aangifteprocedure bij de verzekering zal starten. Deze zal, indien zij het nodig acht, een expert aanstellen om een oordeel uit te spreken over het verband tussen uw gezondheidsklachten en de studie.

In het geval van onenigheid met de arts-onderzoeker of met de door de verzekeringsmaatschappij aangestelde expert, en steeds wanneer u dit nodig acht, kunnen u of in geval van overlijden uw rechthebbenden de verzekeraarmakelaar rechtstreeks in België dagvaarden (Vanbreda Risk & Benefits NV, Plantin en Moretuslei 297, 2140 Antwerpen).

De wet voorziet dat de dagvaarding van de verzekeraar kan gebeuren ofwel voor de rechter van de plaats waar de schade verwekkende feiten zich hebben voorgedaan, ofwel voor de rechter van uw woonplaats, ofwel voor de rechter van de zetel van de verzekeraar.